CLINICAL TRIAL: NCT04146493
Title: Heparin-binding Protein and Heparins
Acronym: HepHep
Status: Completed | Type: Observational
Sponsor: Halla Halldorsdottir (Other)
Collaborators: Karolinska Institutet (Other)
Responsible Party: Sponsor-Investigator, Halla Halldorsdottir, MD, Karolinska University Hospital
Organization: Karolinska University Hospital (Other)
Other Study IDs: 4-2957/2017
Record Dates: First submitted 2019-10-23; First posted 2019-10-31 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Vascular Disease, Peripheral; Thromboprophylaxis; Cardiovascular Diseases
Keywords: Heparin-binding protein; Heparin; Biomarker
MeSH Terms: conditions — Peripheral Vascular Diseases; Cardiovascular Diseases | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Plasma which could theoretically contain DNA
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Vascular surgery group: Patients which are given unfractionated heparin during their vascular surgery.
  Interventions: Diagnostic Test: Blood samples for Heparin-binding protein measurement
- Thromboprophylaxis group: Patients which are given low molecular heparins as a thrombosprofylax after major surgery
  Interventions: Diagnostic Test: Blood samples for Heparin-binding protein measurement
- Cardiothoracic surgery: Patients which are given high dose unfractionated heparin during their open heart surgey
  Interventions: Diagnostic Test: Blood samples for Heparin-binding protein measurement

INTERVENTIONS:
Diagnostic Test: Blood samples for Heparin-binding protein measurement — Blood samples before and after given heparin

SUMMARY:
Heparin-Binding protein is a protein from primary and secretory granluae of white blood cells. It is released when white blood cells become activated and has been advocated as a biomarker for sepsis. The aim of this study is to find out if Heparins in clinical doses can change the level of Heparin-binding protein in plasma.

DETAILED DESCRIPTION:
Blood samples are taken from patients before and after Heparins in clinical doses. The effects of heparins on Heparin-binding protein concentration in plasma is measured. This is a small observational study.

ELIGIBILITY:
Inclusion Criteria:

* Planned endovascular treatment of aortic aneurysm or peripheral vascular surgery where unfractionated heparin in >3000 units are given perioperatively
* Planned subcutaneous low molecular weight heparin as a thromboprophylactic treatment after major surgery or on Intensive Care treated patients.
* Planned open heart surgery with cardiopulmonary bypass.

Exclusion Criteria:

* Under 18 years
* Unable to get informed consent from patient or relative

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A) Patients operated for peripheral vascular disease or aortic disease B) Patients operated for major surgery C) Patients operated for open heart surgery with cardiopulmonary bypass.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2021-11-30 (Actual)

PRIMARY OUTCOMES:
Changes in the level of Heparin-binding protein | Repeated blood sampling during minimum of 1 hour and maximum of 5 hours after given heparin
  Blood samples are taken before and after given heparin

CONTACTS AND LOCATIONS:
Overall Officials: Halla Halldorsdottir, MD, Principal Investigator — Karolinska Institutet
Locations (1):
- Halla Halldorsdottir, Stockholm, Solna, Sweden

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Halldorsdottir H, Lindbom L, Ebberyd A, Oldner A, Weitzberg E. The effect of heparins on plasma concentration of heparin-binding protein: a pilot study. BJA Open. 2024 Jan 27;9:100256. doi: 10.1016/j.bjao.2023.100256. eCollection 2024 Mar. PMID 38318270